CLINICAL TRIAL: NCT02694744
Title: The Effect of Food: An Open-Label, Randomized, Parallel Group Phase 4 Study of the Efficacy and Safety of Patiromer for Oral Suspension With or Without Food for the Treatment of Hyperkalemia (TOURMALINE)
Brief Title: Patiromer With or Without Food for the Treatment of Hyperkalemia
Acronym: TOURMALINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Relypsa, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLY5016-401
Record Dates: First submitted 2016-02-25; First posted 2016-02-29 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Hyperkalemia
Keywords: Treatment of Hyperkalemia; Hyperkalemia; Potassium; Chronic Kidney Disease
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic | interventions — patiromer; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 - Dosing Without Food (Experimental): Patiromer dosing without food
  Interventions: Drug: patiromer
- Group 2 - Dosing With Food (Active Comparator): Patiromer dosing with food
  Interventions: Drug: patiromer

INTERVENTIONS:
Drug: patiromer — 8.4 g/day starting dose, administered orally
  Other Names: Veltassa; RLY5016 for Oral Suspension

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of patiromer administered once daily (QD) when given with food compared to without food (experimental treatment group) for the treatment of hyperkalemia (high potassium in the blood).

DETAILED DESCRIPTION:
Approximately 110 eligible participants with hyperkalemia will be randomly assigned to receive a patiromer starting dose of 8.4- g/day, either with or without food.

All participants will undergo a screening period (1 day) to determine eligibility for study entry. Eligible participants will be treated for 4 weeks and followed for 2 weeks after completing the patiromer treatment. There are six planned clinic visits during the Treatment Period and two planned visits after the last dose of patiromer during the Follow-up Period.

The dose of patiromer may be increased or decreased (titrated) based on participants' individual potassium response.

ELIGIBILITY:
Key Inclusion Criteria:

* Potassium concentration > 5.0 mEq/L from two blood draws at Screening
* Stable RAASi medication, if taking
* Medications taken on a chronic basis are given once daily or twice daily
* Informed consent given

Key Exclusion Criteria:

* Expected need for dialysis
* Major organ transplant
* History of conditions associated with pseudohyperkalemia
* History of swallowing disorder, gastroparesis, bariatric surgery, bowel obstruction or severe gastrointestinal disorders or major gastrointestinal surgery
* Cancer or unstable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director or VP Clinical Development, Study Director — Relypsa, Inc.
Locations (29):
- United States (29):
  - Investigator Site 12, Fountain Valley, California
  - Investigator Site 11, Huntington Beach, California
  - Investigator Site 38, Palm Springs, California
  - Investigator Site 20, Riverside, California
  - Investigator Site 21, San Dimas, California
  - Investigator Site 24, Denver, Colorado
  - Investigator Site 30, Edgewater, Florida
  - Investigator Site 10, Hialeah, Florida
  - Investigator Site 13, Hollywood, Florida
  - Investigator Site 17, Lauderdale Lakes, Florida
  - Investigator Site 16, Lauderdale Lakes, Florida
  - Investigator Site 15, Miami, Florida
  - Investigator Site 43, Miami, Florida
  - Investigator Site 18, Pembroke Pines, Florida
  - Investigator Site 27, Tampa, Florida
  - Investigator Site 44, Meridian, Idaho
  - Investigator Site 39, Aurora, Illinois
  - Investigator Site 23, Flint, Michigan
  - Investigator Site 34, Kansas City, Missouri
  - Investigator Site 41, Las Vegas, Nevada
  - Investigator Site 37, Flushing, New York
  - Investigator Site 36, Norman, Oklahoma
  - Investigator Site 40, Jackson, Tennessee
  - Investigator Site 33, Dallas, Texas
  - Investigator Site 26, San Antonio, Texas
  - Investigator Site 29, San Antonio, Texas
  - Investigator Site 28, San Antonio, Texas
  - Investigator Site 25, San Antonio, Texas
  - Investigator Site 22, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 - Dosing Without Food | Group 2 - Dosing With Food
Started | 57 | 57
Safety Population (Safety Population: All subjects who have taken at least one dose of patiromer.) | 57 | 56
ITT (Two randomized participates from Group 2 were excluded from the analyses for the ITT population.) | 57 | 55
Completed | 51 | 52
Not Completed | 6 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Taking potassium supplement: exclusion 6 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population for analysis included all subjects who were randomized and had taken at least one dose of patiromer.
Groups:
- Group 2 - Dosing With Food: Patiromer dosing with food
  patiromer: 8.4 g/day starting dose, administered orally
  *Note: Two randomized participants in Group 2 -Dosing With Food were excluded from the analyses for the intent-to-treat (ITT) population. One participant who did not receive any patiromer dose. Another participant had an important protocol violation and had no post-baseline serum K+, and was excluded from ITT prior to unblinding.
- Total: Total of all reporting groups
Arm/Group | Group 1 - Dosing Without Food | Group 2 - Dosing With Food | Total
Number analyzed (Participants) | 57 | 55 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 38 | 35 | 73
Age, Continuous [Median (Full Range); unit: years] | 69 [26 to 89] | 66 [48 to 94] | 67 [26 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 40 | 33 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 30 | 63
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 48 | 44 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 57 | 55 | 112

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Serum Potassium in the Target Range (3.8 - 5.0 mEq/L) at Either Week 3 or Week 4
Time Frame: 21 to 28 Days
Population: The intent-to-treat (ITT) population for efficacy analyses includes all subjects who have been randomized and have taken at least one dose of patiromer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 - Dosing Without Food | Group 2 - Dosing With Food
Number analyzed (Participants) | 57 | 55
percentage of participants | 82.5 [70.1 to 91.3] | 87.3 [75.5 to 94.7]
Statistical Analysis 1: Comparison: Group 1 - Dosing Without Food vs Group 2 - Dosing With Food; Test type: Other; If the 95% confidence interval for the w/out food Arm overlapped the confidence interval for the w/ food Arm, the study will conclude that there is no evidence of a statistically significant difference between treatment arms

2. Secondary Outcome: Mean Change in Serum Potassium From Baseline to Week 4
Description: An ANCOVA model was used to estimate the mean serum potassium change from Baseline to Week 4 with baseline serum potassium as a covariate and treatment group, race (white vs all others), and history of Type 1 or 2 diabetes mellitus (yes or no) as factors in the model.
Time Frame: Baseline to Day 28
Population: Only intent-to-treat subjects who were available at both Baseline and Week 4 visits.
Measure: Least Squares Mean (Standard Error); unit: mEq/L
Groups:
- Group 1: Patiromer without Food
- Group 2: Patiromer with Food
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 51 | 49
mEq/L | -0.62 (0.094) | -0.65 (0.088)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Estimation of mean change in serum potassium from Baseline to week 4; Test type: Superiority; p = 0.7893, ANCOVA; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.17 to 0.22]

ADVERSE EVENTS:
Time Frame: Beginning from the time the subject signs the informed consent form until the subject's last study visit, up to 6 weeks.
Description: Treatment emergets AEs (TEAEs) and SAEs were coded in accordance with MedDRA version (18.1). A TEAE is defined as any AE that newly appeared or worsened in severity following initiation of study drug administration.
Groups:
- Group 2 - Dosing With Food: Patiromer dosing with food
  patiromer: 8.4 g/day starting dose, administered orally
  *Note - One randomized participant was excluded from the analysis as this participant did not receive any patiromer dose.
Arm/Group | Group 1 - Dosing Without Food | Group 2 - Dosing With Food
All-Cause Mortality (participants affected / at risk) | 1/57 | 0/56
Serious Adverse Events (participants affected / at risk) | 4/57 | 1/56
Other Adverse Events (participants affected / at risk) | 4/57 | 8/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Dosing Without Food (N=57) | Group 2 - Dosing With Food (N=56)
Angina pectoris (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 - Dosing Without Food (N=57) | Group 2 - Dosing With Food (N=56)
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Headache (Nervous system disorders) | 0 | 3
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements generally provide that PI cannot publish single site data before publication of the multi-site publication, unless 1 year has elapsed since completion of the study at all sites. Thereafter, PI may publish provided that PI shall: provide a copy of the publication to sponsor at least 60 days in advance of submission for publication; delete sponsor's confidential information as requested; and delay publication up to an additional 90 days to permit protection of intellectual property.